CLINICAL TRIAL: NCT01914666
Title: Phase 3 Clinical Study of Duloxetine Hydrochloride in Patients With CLBP - Open Label Long Term Extension Study
Brief Title: An Open Label Extension Study of Duloxetine (LY248686) in Participants With Chronic Low Back Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Shionogi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14949; F1J-JE-HMHC (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-07-31; First posted 2013-08-02 (Estimated); Results first posted 2016-01-27 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2015-12

CONDITIONS: Back Pain Lower Back Chronic
Keywords: Chronic Low Back Pain; CLBP
MeSH Terms: interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Duloxetine (Experimental): Duloxetine 20 milligram (mg) for first week, 40 mg for second week and 60 mg for next 48 weeks administered orally once daily. Tapering week doses of 40 mg for first week and 20 mg for second week.
  Interventions: Drug: Duloxetine

INTERVENTIONS:
Drug: Duloxetine — Administered orally
  Other Names: Cymbalta; LY248686

SUMMARY:
The purpose of the study is to assess the long term safety of duloxetine in participants with Chronic Low Back Pain (CLBP).

ELIGIBILITY:
Inclusion Criteria:

(Consecutive Participants):

* Participants who have completed the 15-week administration in the phase 3 clinical study of Duloxetine hydrochloride in participants with CLBP, study HMGY (NCT01855919)
* Female participants having child-bearing potential must test negative (-) on a pregnancy test

(New Participants):

* Participants with CLBP present for the preceding 6 months or longer
* Participants used nonsteroidal anti-inflammatory drugs for CLBP for less than 14 days on average per month in the past 3 months and less than 14 days in one month prior to study
* Participants having a score of ≥4 on Brief Pain Inventory (BPI) average pain score at participation of study
* Female participants having child-bearing potential must test negative (-) on a pregnancy test

Exclusion Criteria:

(Consecutive Participants):

* Participants having serious or unstable cardiovascular, hepatic, renal, metabolic, respiratory, or hematologic illness, symptomatic peripheral vascular disease, or other medical condition or psychiatric conditions that, in the opinion of investigator, would compromise participation or be likely to lead to hospitalization during the course of the study
* Participants having alanine aminotransferase or aspartate aminotransferase higher than 100 International Units per Liter (IU/L) or total bilirubin higher than 1.6 milligram per deciliter (mg/dL)
* Participants having serum creatinine level higher than 2.0 mg/dL, or had renal transplantation or receiving renal dialysis
* Participants having diagnosis seronegative spondyloarthropathy or rheumatoid arthritis
* Participants having primary painful condition due to other than CLBP
* Participants having uncorrected thyroid disease, uncontrolled narrow-angle glaucoma, history of uncontrolled seizures, or uncontrolled or poorly controlled hypertension
* Participants treating with a monoamine oxidase inhibitor (MAOI) within 14 days or the potential need to use an MAOI during the study or within 5 days of discontinuation of study drug
* Participants answering "yes" to any of the questions about active suicidal ideation/intent/behaviors occurring within the past month (Columbia Suicide Severity Rating Scale, Suicide Ideation section - Questions 4 and 5; Suicidal Behavior section)
* Pregnant participants or participants who are breast-feeding, or wished to be pregnant during the clinical trial period
* Participants cannot use appropriate contraceptive method or do not want to use that from participation of study until one month after the end of administration of the investigational drug
* Participants being considered as inappropriate for participation to the study for any medical or other reason as judged by the investigator

(New Participants):

* Participants having serious or unstable cardiovascular, hepatic, renal, metabolic, respiratory, or hematologic illness, symptomatic peripheral vascular disease, or other medical condition or psychiatric conditions that, in the opinion of investigator, would compromise participation or be likely to lead to hospitalization during the course of the study
* Participants having alanine aminotransferase or aspartate aminotransferase higher than 100 IU/L or total bilirubin higher than 1.6 mg/dL
* Participants having serum creatinine level higher than 2.0 mg/dL, or had renal transplantation or receiving renal dialysis
* Participants having diagnosis seronegative spondyloarthropathy or rheumatoid arthritis
* Participants having primary painful condition due to other than CLBP
* Participants having a history of low back surgery
* Participants having any previous diagnosis of psychosis, bipolar disorder, or schizoaffective disorder
* Participants having major depressive disorder as determined using depression module of the Mini-International Neuropsychiatric Interview
* Participants having uncorrected thyroid disease, uncontrolled narrow-angle glaucoma, history of uncontrolled seizures, or uncontrolled or poorly controlled hypertension
* Participants treating with a MAOI within 14 days or the potential need to use an MAOI during the study or within 5 days of discontinuation of study drug
* Participants answering "yes" to any of the questions about active suicidal ideation/intent/behaviors occurring within the past month (Columbia Suicide Severity Rating Scale, Suicide Ideation section - Questions 4 and 5; Suicidal Behavior section)
* Participants have known hypersensitivity to multiple medications
* Participants are non-ambulatory or require the use of crutches or a walker
* Participants having a history of substance abuse or dependence within the past year, excluding nicotine and caffeine
* Participants having a positive urine drug screen for any substances of abuse
* Participants have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication
* Participants have had previous exposure to duloxetine or completed / withdrawn from any study investigating duloxetine
* Pregnant participants or participants who are breast-feeding, or wished to be pregnant during the clinical trial period
* Participants cannot use appropriate contraceptive method or do not want to use that from participation of study until one month after the end of administration of the investigational drug
* Participants being considered as inappropriate for participation to the study for any medical or other reason as judged by the investigator

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2013-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559 ) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saitama, Japan

RESULTS

PARTICIPANT FLOW:
Groups:
- Naïve: New participants (Pts) administered duloxetine 20 mg during Week 1, 40 mg during Week 2, and 60 mg for Weeks 3-50. Tapering doses of 40 mg for Week 51 and 20 mg for Week 52.
- Rollover (Pre-Placebo): Consecutive participants (randomized to placebo in study F1J-JE-HMGY [NCT#01855919]) administered duloxetine 20 mg during Week 1, 40 mg during Week 2, and 60 mg for Weeks 3-50. Tapering doses of 40 mg for Week 51 and 20 mg for Week 52.
- Rollover (Pre-Duloxetine 60 mg): Consecutive participants (randomized to duloxetine in study F1J-JE-HMGY) administered duloxetine 20 mg during Week 1, 40 mg during Week 2, and 60 mg for Weeks 3-50. Tapering doses of 40 mg for Week 51 and 20 mg for Week 52.
Period: Treatment Period
Arm/Group | Naïve | Rollover (Pre-Placebo) | Rollover (Pre-Duloxetine 60 mg)
Started | 68 | 42 | 41
Received at Least 1 Dose of Study Drug | 68 | 42 | 41
Completed | 55 | 36 | 33
Not Completed | 13 | 6 | 8
Not completed — Lack of Efficacy | 0 | 0 | 2
Not completed — Adverse Event | 10 | 4 | 2
Not completed — Withdrawal by Subject | 3 | 2 | 2
Not completed — Physician Decision | 0 | 0 | 2
Period: Tapering Period
Arm/Group | Naïve | Rollover (Pre-Placebo) | Rollover (Pre-Duloxetine 60 mg)
Started | 59 (4 Pts who discontinued, and 55 Pts who completed Treatment Period entered Tapering Period.) | 39 (3 Pts who discontinued, and 36 Pts who completed Treatment Period entered Tapering Period.) | 40 (7 Pts who discontinued, and 33 Pts who completed Treatment Period entered Tapering Period.)
Completed | 59 | 39 | 40
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) is defined as all randomized participants who received at least 1 dose of study drug, had at least 1 post-dose BPI Pain Severity (average pain) scores. 1 Naïve group participant (pt) received at least 1 dose of study drug but had no post-dose data, was not included in FAS.
Groups:
- Naïve: New participants administered duloxetine 20 milligrams (mg) during Week 1, 40 mg during Week 2, and 60 mg for Weeks 3-50. Tapering doses of 40 mg for Week 51 and 20 mg for Week 52.
- Rollover (Pre-Placebo): Consecutive participants (randomized to placebo in study F1J-JE-HMGY) administered duloxetine 20 mg during Week 1, 40 mg during Week 2, and 60 mg for Weeks 3-50. Tapering doses of 40 mg for Week 51 and 20 mg for Week 52.
- Total: Total of all reporting groups
Arm/Group | Naïve | Rollover (Pre-Placebo) | Rollover (Pre-Duloxetine 60 mg) | Total
Number analyzed (Participants) | 67 | 42 | 41 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.3 (13.9) | 57.6 (12.0) | 58.8 (11.1) | 56.4 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 22 | 22 | 80
  Male | 31 | 20 | 19 | 70
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 67 | 42 | 41 | 150
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Japan | 67 | 42 | 41 | 150

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Drug Related Adverse Events (AEs) or Any Serious AE's
Description: A summary of serious AEs and all other non-serious AEs, regardless of causality, is located in the Reported Adverse Event module.
Time Frame: Week 53
Population: All the enrolled participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Naïve | Rollover (Pre-Placebo) | Rollover (Pre-Duloxetine 60 mg)
Number analyzed (Participants) | 68 | 42 | 41
participants
  Drug Related AEs | 42 | 16 | 18
  Serious AEs | 4 | 3 | 1

2. Secondary Outcome: Change From Baseline in Brief Pain Inventory (BPI) Pain Severity Item and Interference Item to Week 50
Description: A self-reported scale measuring severity of pain and interference on function. Severity scores: 0 (no pain) to 10 (severe pain) on each question assessing worst pain, least pain, and average pain in past 24 hours, and pain right now. Interference scores: 0 (does not interfere) to 10 (completely interferes) on each question assessing interference of pain in past 24 hours for general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life. Average interference = average of non-missing scores of individual interference items.
Time Frame: Baseline, Week 50
Population: (FAS): All randomized participants who received at least 1 dose of study drug and had at least 1 post-dose BPI pain severity (average pain) scores. The last observation carried forward (LOCF) was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Naïve | Rollover (Pre-Placebo) | Rollover (Pre-Duloxetine 60 mg)
Number analyzed (Participants) | 67 | 42 | 41
units on a scale
  Average Pain | -3.30 (1.45) | -3.79 (1.66) | -2.88 (1.81)
  Worst Pain | -4.16 (1.91) | -4.71 (2.21) | -3.24 (1.88)
  Least Pain | -1.82 (1.54) | -2.52 (1.77) | -2.12 (1.71)
  Pain Right Now | -2.70 (1.87) | -3.93 (1.74) | -2.68 (1.90)
  General Activity | -3.22 (2.30) | -3.26 (2.51) | -2.24 (2.75)
  Mood | -2.52 (2.55) | -3.12 (2.37) | -2.07 (2.49)
  Walking Ability | -2.09 (2.16) | -2.74 (2.26) | -1.71 (3.11)
  Normal Work | -3.22 (2.49) | -3.21 (2.23) | -2.05 (2.78)
  Relationship with People | -1.42 (2.15) | -1.79 (2.37) | -0.83 (1.82)
  Sleep | -1.73 (2.12) | -2.40 (2.56) | -1.34 (2.22)
  Enjoyment of Life | -2.07 (2.27) | -2.50 (2.55) | -1.83 (2.40)
  Average of 7 Interference Items | -2.33 (1.81) | -2.72 (2.05) | -1.72 (2.21)

3. Secondary Outcome: Patient Global Impression of Improvement (PGI-Improvement) to Week 50
Description: PGI-I measures a participant's perception of improvement at the time of assessment compared with the start of treatment. Score ranges from 1 (very much better) to 7 (very much worse).
Time Frame: Week 50
Population: FAS: All randomized participants who received at least 1 dose of study drug and had at least 1 post-dose BPI pain severity (average pain) scores. LOCF was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Naïve | Rollover (Pre-Placebo) | Rollover (Pre-Duloxetine 60 mg)
Number analyzed (Participants) | 67 | 42 | 41
units on a scale | 2.12 (0.88) | 2.05 (0.82) | 2.61 (1.16)

4. Secondary Outcome: Change From Baseline in Clinical Global Impression of Severity (CGI-Severity) to Week 50
Description: CGI-S measures severity of illness at the time of assessment compared with start of treatment with scores ranging from 1 (normal, not at all ill) to 7 (among the most extremely ill participants).
Time Frame: Baseline, Week 50
Population: FAS: All randomized participants who received at least 1 dose of study drug and had at least 1 post-dose BPI pain severity (average pain) score. LOCF was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Naïve | Rollover (Pre-Placebo) | Rollover (Pre-Duloxetine 60 mg)
Number analyzed (Participants) | 67 | 42 | 41
units on a scale | 2.09 (0.81) | 2.00 (0.73) | 2.73 (0.98)

5. Secondary Outcome: Change From Baseline in Roland Morris Disability Questionnaire (RMDQ-24) to Week 50
Description: RMDQ-24 is a participant completed questionnaire and measures the degree of disability due to back pain. The questionnaire consists of 24 statements and the participant was instructed to put a mark next to each appropriate statement. The number of statements marked was summed by the clinician for a total score. The total score ranged from 0 (no disability) to 24 (severe disability).
Time Frame: Baseline, Week 50
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Naïve | Rollover (Pre-Placebo) | Rollover (Pre-Duloxetine 60 mg)
Number analyzed (Participants) | 67 | 42 | 41
units on a scale | -3.69 (3.76) | -5.50 (5.64) | -3.29 (4.56)

6. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) to Week 50
Description: SF-36 Health Status Survey is a generic, health-related scale assessing participant's quality of life on 8 domains: physical functioning, social functioning, bodily pain, vitality, mental health, role-physical, role-emotional and general health. Each domain is scored by summing the individual items and transforming the scores into a 0 to 100 scale, with higher scores indicating better health status or functioning.
Time Frame: Baseline, Week 50
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Naïve | Rollover (Pre-Placebo) | Rollover (Pre-Duloxetine 60 mg)
Number analyzed (Participants) | 67 | 42 | 41
units on a scale
  Physical Functioning | 10.60 (15.21) | 9.52 (21.91) | 10.12 (17.66)
  Role (Physical) | 16.88 (20.73) | 11.31 (24.24) | 7.01 (21.66)
  Bodily Pain | 17.64 (16.32) | 20.26 (22.09) | 12.62 (16.58)
  General Health | 8.42 (13.81) | 8.90 (14.54) | 5.51 (18.57)
  Vitality | 10.07 (16.64) | 13.24 (23.15) | 6.10 (18.93)
  Social Functioning | 6.90 (21.24) | 8.63 (19.22) | 3.35 (20.16)
  Role (Emotional) | 11.57 (20.05) | 11.51 (23.20) | 4.47 (16.99)
  Mental Health | 5.97 (15.31) | 8.81 (14.89) | 4.63 (14.12)

7. Secondary Outcome: Change From Baseline in European Quality of Life Questionnaire-5 Dimension (EQ-5D) to Week 50
Description: The EQ-5D is a generic, multidimensional, health-related, quality-of-life instrument. The profile allows participants to rate their health state in 5 health domains: mobility, self-care, usual activities, pain/discomfort, and mood using a three level scale (no problem, some problems, and major problems). These combinations of attributes were converted into a weighted health-state Index Score according to the Japan population-based algorithm ranging from -0.111 to 1.0, with higher scores indicating better quality of life.
Time Frame: Baseline, Week 50
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Naïve | Rollover (Pre-Placebo) | Rollover (Pre-Duloxetine 60 mg)
Number analyzed (Participants) | 67 | 42 | 41
units on a scale | 0.16 (0.16) | 0.15 (0.15) | 0.11 (0.15)

8. Secondary Outcome: Change From Baseline in Beck Depression Inventory-II (BDI-II) to Week 50
Description: BDI-II is a 21-item, participant-completed questionnaire to assess characteristics of depression. Each of the 21 items corresponding to symptoms of depression were scored on a 4-point scale ranging from 0 to 3 and was summed to give a single score. A total score of 0-13 was considered minimal range, 14-19 was mild, 20-28 was moderate, and 29-63 was severe.
Time Frame: Baseline, Week 50
Population: FAS: All randomized participants who received at least 1 dose of study drug and had baseline and at least 1 post-dose BPI pain severity (average pain) scores. LOCF was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Naïve | Rollover (Pre-Placebo) | Rollover (Pre-Duloxetine 60 mg)
Number analyzed (Participants) | 67 | 42 | 41
units on a scale | -1.81 (5.32) | -1.83 (5.00) | -0.56 (3.75)

9. Secondary Outcome: Change From Baseline in Columbia Suicide Severity Rating Scale (C-SSRS) to Week 52
Description: C-SSRS captures occurrence, severity, and frequency of suicide-related thoughts and behaviors. Suicidal behavior is defined as a "yes" answer to any of 5 suicidal behavior questions: preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, and completed suicide. Suicidal ideation is defined as a "yes" answer to any one of 5 suicidal ideation questions: wish to be dead, and 4 different categories of active suicidal ideation.
Time Frame: Baseline, Week 53
Population: All randomized participants who received at least 1 dose of study drug, responded no at baseline to the suicide related questionnaire and had data at post-treatment for each question.LOCF was used.
Measure: Number; unit: participants
Arm/Group | Naïve | Rollover (Pre-Placebo) | Rollover (Pre-Duloxetine 60 mg)
Number analyzed (Participants) | 65 | 39 | 40
participants
  Suicidal Ideation- wish to be dead (n=65,39,40) | 0 | 0 | 0
  Nonspecific suicidal thoughts (n=67,42,41) | 0 | 0 | 0
  Suicidal Behavior (n=67,42,41) | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With Fall Events From Fall Questionnaire
Description: Participants evaluated their experience with and details of falls which were recorded. Percentage = (number of participants with fall events) /(total in treatment group) * 100.
Time Frame: Week 53
Population: All the enrolled participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Naïve | Rollover (Pre-Placebo) | Rollover (Pre-Duloxetine 60 mg)
Number analyzed (Participants) | 68 | 42 | 41
participants | 13 | 5 | 6

ADVERSE EVENTS:
Description: AEs for all participants who received at least one dose of study drug.
Groups:
- Naïve, Rollover (Pre-Placebo), Rollover (Pre-Duloxetine 60 mg): All participants from Naïve, Rollover (Pre-Placebo), Rollover (Pre-Duloxetine 60 mg) groups combined.
Arm/Group | Naïve, Rollover (Pre-Placebo), Rollover (Pre-Duloxetine 60 mg)
Serious Adverse Events (participants affected / at risk) | 8/151
Other Adverse Events (participants affected / at risk) | 129/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naïve, Rollover (Pre-Placebo), Rollover (Pre-Duloxetine 60 mg) (N=151)
Angle closure glaucoma (Eye disorders) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 1 (1)
Death (General disorders) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Brain stem infarction (Nervous system disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Naïve, Rollover (Pre-Placebo), Rollover (Pre-Duloxetine 60 mg) (N=151)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 3 (4)
Tinnitus (Ear and labyrinth disorders) | 5 (5)
Vertigo (Ear and labyrinth disorders) | 4 (4)
Chalazion (Eye disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (1)
Retinal haemorrhage (Eye disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 7 (7)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3)
Anal fissure (Gastrointestinal disorders) | 1 (1)
Aphthous stomatitis (Gastrointestinal disorders) | 1 (1)
Barrett's oesophagus (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 15 (15)
Dental caries (Gastrointestinal disorders) | 8 (8)
Diarrhoea (Gastrointestinal disorders) | 4 (4)
Dyschezia (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Gastric polyps (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 16 (18)
Periodontal disease (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Chest discomfort (General disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Feeling abnormal (General disorders) | 2 (2)
Malaise (General disorders) | 4 (4)
Oedema peripheral (General disorders) | 1 (1)
Thirst (General disorders) | 9 (9)
Hepatic mass (Hepatobiliary disorders) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 2 (2)
Sarcoidosis (Immune system disorders) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1)
Acarodermatitis (Infections and infestations) | 2 (2)
Acute tonsillitis (Infections and infestations) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 6 (7)
Cystitis (Infections and infestations) | 2 (3)
Erythema infectiosum (Infections and infestations) | 1 (1)
Furuncle (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 5 (6)
Gingival abscess (Infections and infestations) | 1 (1)
Gingival infection (Infections and infestations) | 2 (2)
Gingivitis (Infections and infestations) | 2 (3)
Herpes zoster (Infections and infestations) | 1 (1)
Infected dermal cyst (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 7 (7)
Nasopharyngitis (Infections and infestations) | 37 (48)
Oral herpes (Infections and infestations) | 1 (1)
Paronychia (Infections and infestations) | 1 (1)
Periodontitis (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 5 (5)
Pneumonia (Infections and infestations) | 2 (2)
Subcutaneous abscess (Infections and infestations) | 1 (2)
Tonsillitis (Infections and infestations) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 1 (1)
Bone contusion (Injury, poisoning and procedural complications) | 4 (4)
Burns first degree (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 17 (26)
Epicondylitis (Injury, poisoning and procedural complications) | 5 (5)
Excoriation (Injury, poisoning and procedural complications) | 2 (2)
Hand fracture (Injury, poisoning and procedural complications) | 2 (2)
Heat illness (Injury, poisoning and procedural complications) | 2 (3)
Laceration (Injury, poisoning and procedural complications) | 1 (1)
Ligament injury (Injury, poisoning and procedural complications) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 8 (12)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1)
Muscle injury (Injury, poisoning and procedural complications) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 2 (2)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 4 (4)
Blood creatine phosphokinase increased (Investigations) | 2 (2)
Blood creatinine increased (Investigations) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 1 (2)
Blood triglycerides increased (Investigations) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 2 (2)
Liver function test abnormal (Investigations) | 4 (4)
Occult blood (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2)
Gout (Metabolism and nutrition disorders) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 (2)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (13)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (6)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 3 (3)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4)
Periarthritis (Musculoskeletal and connective tissue disorders) | 8 (10)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 (2)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 2 (2)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 1 (1)
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Morton's neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Autonomic nervous system imbalance (Nervous system disorders) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1)
Cervical radiculopathy (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 8 (11)
Dizziness postural (Nervous system disorders) | 5 (5)
Dysgeusia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 10 (11)
Hypoaesthesia (Nervous system disorders) | 2 (2)
Intercostal neuralgia (Nervous system disorders) | 1 (1)
Myelopathy (Nervous system disorders) | 1 (1)
Radiculitis cervical (Nervous system disorders) | 1 (1)
Sensory disturbance (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 29 (30)
Syncope (Nervous system disorders) | 1 (1)
Tension headache (Nervous system disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 4 (4)
Dysuria (Renal and urinary disorders) | 2 (2)
Hypertonic bladder (Renal and urinary disorders) | 3 (3)
Pollakiuria (Renal and urinary disorders) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 1/81 (1)
Gynaecomastia (Reproductive system and breast disorders) | 1/70 (1)
Metrorrhagia (Reproductive system and breast disorders) | 1/81 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (4)
Asteatosis (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Skin tightness (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2)
Urticaria cholinergic (Skin and subcutaneous tissue disorders) | 1 (1)
Hot flush (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
Peripheral coldness (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
FAS:all randomized pts who received at least 1 dose of study drug and had at least 1 post-dose BPI pain severity (average pain) score. 1 Naïve group pt received at least 1 dose of study drug but had no post-dose data and not included in FAS.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days